CLINICAL TRIAL: NCT06240884
Title: Comparison of Ultrasound-guided Infraspinatus Tubercle Muscle (ITM) Interfascial Block and Interosseous Groove Nerve Block (ISB) for Postoperative Pain Management After Shoulder Arthroscopy: a Randomised, Non-inferiority Study
Brief Title: Postoperative Analgesic Effect of Infraspinatus-teres Minor Inter-fascial Block in Patients Undergoing Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, professor, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KY-676
Record Dates: First submitted 2024-01-02; First posted 2024-02-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Pain
Keywords: Infraspinatus-teres minor (ITM) interfascial block; shoulder arthroscopy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infraspinatus-teres minor interfascial block (Experimental): Patients will receive Infraspinatus-teres Minor Interfascial Block with 20 ml of 0.375% ropivacaine prior to induction of general anesthesia.
  Interventions: Procedure: Infraspinatus-teres minor interfascial block
- interscalene block (Active Comparator): The patient underwent an ultrasound-guided brachial plexus nerve block in the interosseous sulcus using 20 ml of 0.375% ropivacaine.
  Interventions: Procedure: interscalene block

INTERVENTIONS:
Procedure: Infraspinatus-teres minor interfascial block — After identifying the infraspinatus and teres minor muscles on the posterior surface of the scapular neck. Under real-time ultrasound guidance, the needle is advanced into the interfascial plane between the infraspinatus and teres minor muscles using an in-plane technique, and after confirming the fascial opening with 3 to 5 mL of 0.375% ropivacaine (20 mL total dose), the remaining 0.375% ropivacaine is injected. After extubation and the patients were awake, anesthesiologists who were unaware of the study subgroups began to assess the analgesic effect of the patients' block at rest using the numeric pain rating scale (NRS) at 0.5h, 3h, 6h, 12h, 18h, 24h, and 48h postoperatively.
  Arms: Infraspinatus-teres minor interfascial block
Procedure: interscalene block — The tip of the needle was placed between the C5 and C6 nerve roots, and after a bloodless retraction with 0.5 to 1 ml of 0.375% ropivacaine to confirm nerve displacement, the remaining 0.375% ropivacaine was injected (total dose of 20 ml). Subsequently, the catheter was inserted over the needle and the needle was withdrawn.After extubation and the patients were awake, anesthesiologists who were unaware of the study subgroups began to assess the analgesic effect of the patients' block at rest using the numeric pain rating scale (NRS) at 0.5h, 3h, 6h, 12h, 18h, 24h, and 48h postoperatively.
  Arms: interscalene block

SUMMARY:
It is proposed to investigate the effectiveness of ultrasound-guided intertrochanteric block of the infraspinatus minor round myofascial block not inferior to the interosseous groove brachial plexus nerve block in postoperative analgesia and overall quality of recovery in shoulder surgery.

DETAILED DESCRIPTION:
Intersulcus brachial plexus nerve block is considered to be the best method for pain nerve block after shoulder joint surgery. It can not only effectively reduce the postoperative pain and discomfort of patients, but also reduce the intraoperative demand for opioids. However, the use of intermuscular brachial plexus block should be prohibited when the patient has a clotting disorder or is taking anticoagulant drugs, has a local infection or a systemic infection. There may also be anesthesia risks such as nerve damage, vascular damage, respiratory depression, and diaphragmatic paralysis with dyspnea.

Infraspinatus-teres minor (ITM), first proposed by Shin Hyung Kim, is a single-site injection in the interfascial plane between Infraspinatus and teres minor. Once the IS and Tm on the humeral head area are identified, by moving the probe mediocaudally, the interfascial structure of the IS and Tm can be traced along the glenohumeral joint, scapular neck area. On autopsy, local anesthetics were found to have spread to the suprascapular and axillary nerves. This result suggests that interfascia block injection of local anesthetics between the infraspinatus and teres minor muscles may help relieve pain in the upper shoulder, back, and external sensory areas. At present, there are few clinical reports on the use of infraspinatus-teres minor interfascial block for postoperative analgesia of shoulder joint, and the postoperative analgesia effect is only reported in individual cases, without comparison with other nerve blocks There are few studies on the clinical application of ITM block, but ISB has become the best method for postoperative analgesia of shoulder joint surgery. the investigators designed a prospective, randomized controlled, non-inferior study to investigate the efficacy of ultrasound-guided subaspina-teres minor interfascial block in analgesia and overall quality of recovery after shoulder joint surgery.

The primary outcome indicator was the area under the NRS curve at rest in the 0-24h postoperative period

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder joint surgery in Jiaxing First Hospital from November 2023 to February 2024;
2. Age 18-80 years old;
3. ASA Grade I-III;
4. The duration of surgery is expected to be 1-3h

Exclusion Criteria:

1. accompanied by nerve injury or disease around the shoulder joint, including thoracic outlet syndrome, Multiple sclerosis, cervical disc disease with ipsilateral radiculopathy, etc.
2. accompanied by abnormal sensory or motor function of the upper limb;
3. Active infection at the puncture site, or coagulation dysfunction (hemophilia, von willeophilia, or International normalized ratio [INR]>2);
4. Patients with severe respiratory diseases and a serious history of cardiovascular and cerebrovascular diseases;
5. ipsilateral shoulder joint surgery history;
6. Patients with nerve block failure;
7. Allergic to local anesthetics;
8. Long-term use of opioids (duration ≥3 months or duration ≥1 month and daily dose ≥5mg morphine equivalent);
9. Operation time <1h or >3h
10. Patients and their families refused surgical anesthesia and were unable to complete the questionnaire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Area under the NRS curve at rest during 0-24h postoperatively | 0-24 hours after surgery
  Anesthesiologists who were not aware of the study subgroups began to assess the analgesic effect of the patients' block at rest using the numeric pain rating scale (NRS) at 0.5h, 3h, 6h, 12h, 18h, and 24h postoperatively.Score range from 0 (no pain) to 10 (worst pain possible).

SECONDARY OUTCOMES:
Complications | during 48 hours after operation
  number of participants developed complications
Asses The postoperative opioid consumption | 24 hours postoperatively
  the postoperative opioid consumption during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: QINGhe ZHOU, Principal Investigator — deputy chair of board
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
research direction

REFERENCES:
- [Result] Kim SH, Yeo IS, Jang J, Jung HE, Chun YM, Yang HM. Infraspinatus-teres minor (ITM) interfascial block: a novel approach for combined suprascapular and axillary nerve block. Reg Anesth Pain Med. 2024 Jan 11;49(1):67-72. doi: 10.1136/rapm-2023-104738. PMID 37491150